CLINICAL TRIAL: NCT03183479
Title: The Effects of Fibrinogen Concentrate Infusion on Perioperative Blood Loss and Allogeneic Blood Conservation in Patients Undergoing Scoliosis Surgery
Brief Title: The Effects of Fibrinogen Concentrate Infusion on Blood Loss and Allogeneic Blood Conservation in Scoliosis Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Weiyun Chen, Principal Investigator, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PUMCH-FC
Record Dates: First submitted 2017-06-05; First posted 2017-06-12 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Scoliosis; Adolescence; Bleeding; Surgery
Keywords: adolescent idiopathic scoliosis; fibrinogen concentrate; perioperative blood loss; transfusion
MeSH Terms: conditions — Scoliosis; Hemorrhage | interventions — Fibrinogen; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: After randomization, the unblinded independent investigator will be in charge of fibrinogen concentrate (drug) or placebo preparation, which will be performed in a laboratory next to the operating room. When the patient meets the inclusion criteria and is enrolled in the study, the functional fibrinogen tests will be done in the same laboratory by the same researcher, and drug or placebo will be prepared in sterile bags with opaque covers afterwards. Fibrinogen concentrate will be diluted in 100mL of sterile water or an equivalent volume of 0.9% saline solution as placebo and will be delivered to the operating room by the investigator. The anesthesiologists, the surgical staff, and the patients will all be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): The patients in treatment group will receive Fibrinogen Concentrate Human administration.
  Interventions: Drug: Fibrinogen Concentrate Human
- Control group (Placebo Comparator): The patients in control group will be administered with normal saline solution as placebo.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Fibrinogen Concentrate Human — After start of surgery when all pedicle screws are placed, the patients in treatment group will receive fibrinogen concentrate 30mg kg-1. For safety concern, functional fibrinogen will be measured and the maximum fibrinogen concentrate administration for each individual shall not exceed 2g. Fibrinogen concentrate will be diluted in 100mL of sterile water and then be administered to patients.
  Other Names: FIBRORAAS
  Arms: Treatment group
Drug: Normal saline — 100mL normal saline will be administered to patients in control group as placebo
  Arms: Control group

SUMMARY:
Allogeneic blood products transfusions are often necessary to treat perioperative bleeding in patients undergoing complex scoliosis surgeries. A prospective, randomized trial is designed to evaluate if the infusion of fibrinogen concentrate may reduce allogeneic blood transfusion in patients undergoing scoliosis surgery. Eligible patients will be randomly assigned to treatment group (fibrinogen concentrate infusion) and control group (normal saline infusion), and functional fibrinogen will be measured to guide the infusion of fibrinogen concentrate. Perioperative blood loss, intraoperative blood loss, and the amount of perioperative allogeneic blood transfusion will be compared between the two groups to determine the effect of fibrinogen concentrate infusion.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blinded, placebo controlled trial to evaluate the effects of fibrinogen concentrate infusion on perioperative blood loss and the amount of perioperative allogeneic blood transfusion in patients undergoing scoliosis surgery.

Recently, the inherent risks of blood, along with the continued rise in blood costs, activated the development and use of alternatives to blood transfusion. Fibrinogen concentrate may limit postoperative bleeding and lead to a significant reduction in allogeneic blood products transfusions in cardiac surgery and craniosynostosis surgery. However, the effect of fibrinogen concentrate in scoliosis surgery is still uncertain. Therefore, a prospective, randomized trial is designed to evaluate if the infusion of fibrinogen concentrate may reduce allogeneic blood transfusion in patients undergoing scoliosis surgery.

Patients older than 12y/o with adolescent idiopathic scoliosis planed for elective posterior scoliosis correction surgery will be enrolled for this study after informed consent. Patients will be randomly assigned to a treatment group or a control group. Functional fibrinogen will be measured using TEG 5000 (Haemoscope Corp, IL, USA) at the start of surgery and the results of FLEV and MA will be recorded. After pedicle screw placement, a second functional fibrinogen will be measured and the patients in treatment group will receive fibrinogen concentrate (FIBRORAAS, Shanghai RAAS Blood Products Co, Ltd, Shanghai, China) 30mg kg-1. For safety concern, the maximum fibrinogen concentrate administration for each individual shall not exceed either 2g. Patients in the control group will receive placebo treatment with normal saline. After 15 minutes from fibrinogen concentrate or placebo administration, a third functional fibrinogen measurement will be performed to assess the effect of treatment. The following treatment will be guaranteed by the standard protocol in the presence of ongoing bleeding.

Data includes all the demographics, preoperative conditions, procedure details, intraoperative data, and outcome measurements will be recorded. Additional data including FLEV and MA value, as well as fibrinogen values both preoperatively and at the arrival at wards. The primary endpoint of this study will be the total perioperative blood loss, and secondary endpoints will include: perioperative blood loss per fused level, intraoperative blood loss per fused level, the amount of postoperative drainage, the amount of postoperative drainage per fused level, total units of perioperative allogeneic pRBCs transfused, total volume of FFP transfused, total PLT units transfused. Safety endpoints will include operative mortality and perioperative thromboembolic complications.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed as adolescent idiopathic scoliosis
* planed for elective posterior scoliosis correction surgery at Peking Union Medical College Hospital

Exclusion Criteria:

* preoperative anemia
* preoperative congenital or acquired coagulopathy
* ongoing anticoagulation therapy or drug intake that could cause bleeding
* clinical signs or diagnosis of acute thromboembolism
* emergency surgery
* redo surgery

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 102 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Perioperative blood loss | hospital stay up to 30 days
  the total amount of intraoperative and postoperative blood loss

SECONDARY OUTCOMES:
Perioperative blood loss per fused level | hospital stay up to 30 days
  amount of intraoperative and postoperative blood loss divided by the number of surgical fused levels
Intraoperative blood loss | From the time of skin incision until wound closure, assessed up to 12 hours
  the amount of intraoperative blood loss
Intraoperative blood loss per fused level | From the time of skin incision until wound closure, assessed up to 12 hour
  amount of intraoperative blood loss divided by the number of surgical fused levels
Postoperative drainage | hospital stay up to 30 days
  the amount of postoperative drainage
Postoperative drainage per fused level | hospital stay up to 30 days
  amount of postoperative drainage divided by the number of surgical fused levels
Perioperative allogeneic red blood cell (RBC) transfusion | hospital stay up to 30 days
  total units of RBC transfused perioperatively
Perioperative plasma transfusion | hospital stay up to 30 days
  total volume of plasma transfused perioperatively
Perioperative platelets transfusion | hospital stay up to 30 days
  total units of platelets transfused perioperatively

CONTACTS AND LOCATIONS:
Overall Officials: Weiyun Chen, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Coded data is anticipated to be shared with potential collaborators.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Anticipated that data from the study will become available within 5 years after publication of main data.
Access Criteria: Data would only be shared with IRB approved collaborators.

REFERENCES:
- [Derived] Chen W, Shen J, Zhang Y, Hu A, Liang J, Ma L, Yu X, Huang Y. A randomised controlled trial of fibrinogen concentrate during scoliosis surgery. Anaesthesia. 2020 Nov;75(11):1476-1481. doi: 10.1111/anae.15124. Epub 2020 Jun 4. PMID 32500569